CLINICAL TRIAL: NCT02758652
Title: Molecular Mechanisms Leading to Chemoresistance in Epithelial Ovarian Cancer
Acronym: CHEMOVA
Status: Active, not recruiting | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other); University of Helsinki (Other)
Responsible Party: Principal Investigator, Annika Auranen, Chief in gynecological oncology, Tampere University Hospital
Other Study IDs: R15134
Record Dates: First submitted 2016-04-05; First posted 2016-05-02 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Ovarian Cancer
Keywords: chemoresistance; miRNA; microRNA
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, urine and tissue samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Epithelial ovarian cancer is the most lethal gynecological malignancy in developed countries and the fifth most common cause of cancer-related death in women. Poor prognosis is due to challenges in early diagnosis and development of inevitable resistance to chemotherapy in majority of patients despite of good initial treatment response. The purpose of this prospective study is to analyze variation in microRNA expression in prediction of primary treatment response and the role of microRNAs in development of chemoresistance in epithelial ovarian cancer.

• Objectives: To screen microRNAs from prospectively collected plasma, urine and tumor samples from patients diagnosed with epithelial ovarian cancer. Samples are analyzed for microRNA expression and differential expression is correlated with primary treatment response, progression-free survival and overall survival.

• Methods: Plasma, urine and tumor samples are collected at primary surgery (open surgery or diagnostic laparoscopy) or interval debulking surgery, at 1st, 3rd and 6th neoadjuvant or adjuvant chemotherapy and at progression for high-throughput screening of microRNA expression by array technology.

DETAILED DESCRIPTION:
Inclusion criteria:

patients operated for a suspected ovarian malignancy in the Department of Obstetrics and Gynecology in Tampere University Informed consent obtained

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age, informed consent.

Exclusion Criteria:

* Informed consent not provided, age under 18 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed epithelial ovarian cancer patients operated inTampere University Hospital, Finland.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2016-05; Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
miRNA expression profile as measured by miRNA array | 5 years
  Expression profile calculated with bioinformatical analysis

SECONDARY OUTCOMES:
Progression-free survival | 5 years
  Time from diagnosis to disease relapse
Over-all survival | 5 years
  Timo from diagnosis to death

CONTACTS AND LOCATIONS:
Overall Officials: Annika Auranen, adj prof, Principal Investigator — Chief of Gynecological Oncology
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Savolainen K, Scaravilli M, Ilvesmaki A, Staff S, Tolonen T, Maenpaa JU, Visakorpi T, Auranen A. Expression of the miR-200 family in tumor tissue, plasma and urine of epithelial ovarian cancer patients in comparison to benign counterparts. BMC Res Notes. 2020 Jul 1;13(1):311. doi: 10.1186/s13104-020-05155-6. PMID 32611374